CLINICAL TRIAL: NCT02413333
Title: Comparison of Two One-Step Hydrogen Peroxide Lens Care Solutions in Symptomatic Contact Lens Wearers
Brief Title: Clear Care® Plus vs. PeroxiClear™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: LCD913-P001
Record Dates: First submitted 2015-04-07; First posted 2015-04-09 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-07

CONDITIONS: Refractive Error
Keywords: Contact lens solution
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clear Care Plus, then PeroxiClear (Other): Clear Care Plus contact lens solution in Period 1, followed by PeroxiClear contact lens solution in Period 2. Each product used daily per packaging instructions with participant's habitual silicone hydrogel contact lenses for approximately 30 cleaning cycles.
  Interventions: Device: Clear Care Plus contact lens solution; Device: PeroxiClear contact lens solution; Device: Silicone hydrogel contact lenses
- PeroxiClear, then Clear Care Plus (Other): PeroxiClear contact lens solution in Period 1, followed by Clear Care Plus contact lens solution in Period 2. Each product used daily per packaging instructions with participant's habitual silicone hydrogel contact lenses for approximately 30 cleaning cycles.
  Interventions: Device: Clear Care Plus contact lens solution; Device: PeroxiClear contact lens solution; Device: Silicone hydrogel contact lenses

INTERVENTIONS:
Device: Clear Care Plus contact lens solution — 3% hydrogen peroxide solution with Hydraglyde Moisture Matrix for cleaning, disinfection and overnight storage of contact lenses
  Other Names: Clear Care Plus
Device: PeroxiClear contact lens solution — 3% hydrogen peroxide solution for cleaning, disinfection and overnight storage of contact lenses
  Other Names: PeroxiClear
Device: Silicone hydrogel contact lenses — 2-week/monthly replacement contact lenses per participant's habitual brand

SUMMARY:
The purpose of this study is to evaluate Clear Care® Plus compared to PeroxiClear™ for mean residual peroxide in used lens cases collected at Day 30 after neutralization at recommended storage time.

DETAILED DESCRIPTION:
Participants will wear habitual lenses on a daily wear basis and use the assigned test solution for daily lens care.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent form;
* Adapted, 2-week/monthly replacement silicone hydrogel contact lens wearers (at least 2 months);
* Willing to wear study lenses daily wear only on a daily basis (7 days per week and at least 4 hours per day) and attend all study visits;
* Symptoms of contact lens related dryness as defined by the Symptomatic Pre-Screening Questionnaire;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Current hydrogen peroxide-based solution user;
* Routinely sleeps in lenses at least 1 night per week over the last 3 months prior to enrollment;
* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear;
* Any systemic diseases that may affect the eye or be exacerbated by use of contact lenses or contact lens solutions or which could prevent wearing lenses at least 4 hours per day;
* Use of systemic or ocular medications for which contact lens wear could be contraindicated;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* History of herpetic keratitis, ocular surgery, or irregular cornea;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Vision Care, Global Medical Affairs, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ten investigational centers located in the United States.
Pre-assignment Details: All randomized participants (132). One enrolled participant discontinued prior to randomization.
Period: Period 1
Arm/Group | Clear Care Plus, Then PeroxiClear | PeroxiClear, Then Clear Care Plus
Started | 66 | 66
Randomized and Treated | 66 | 66
Completed | 65 | 65
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Reason Not Specified | 0 | 1
Period: Period 2
Arm/Group | Clear Care Plus, Then PeroxiClear | PeroxiClear, Then Clear Care Plus
Started | 65 | 65
Completed | 64 | 65
Not Completed | 1 | 0
Not completed — Protocol Deviation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set, defined as all participants randomized and treated. Two participants inadvertently used the incorrect product during the second period, and they are defined according to the treatment received.
Groups:
- Clear Care Plus, Then PeroxiClear: Clear Care Plus was used in Period 1, then PeroxiClear in Period 2.
- PeroxiClear, Then Clear Care Plus: PeroxiClear was used in Period 1, then Clear Care Plus in Period 2.
- Clear Care Plus, Then Clear Care Plus: Clear Care Plus was used in Period 1 and in Period 2.
- PeroxiClear, Then PeroxiClear: PeroxiClear was used in Period 1 and in Period 2.
- Total: Total of all reporting groups
Arm/Group | Clear Care Plus, Then PeroxiClear | PeroxiClear, Then Clear Care Plus | Clear Care Plus, Then Clear Care Plus | PeroxiClear, Then PeroxiClear | Total
Number analyzed (Participants) | 65 | 65 | 1 | 1 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (11.2) | 35.7 (11.8) | 42.0 (NA) — Single data point | 38.0 (NA) — Single data point | 36.7 (11.4)
Age, Customized [Number; unit: participants]
  18-64 years | 65 | 64 | 1 | 1 | 131
  ≥65 years | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 49 | 1 | 1 | 103
  Male | 13 | 16 | 0 | 0 | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Residual Peroxide at Day 30
Description: The used lens case was collected after approximately 30 days of use. Remaining liquid was removed and dry cases were shipped to a lab for analysis. 10 mL of the appropriate solution was added to each collected case. Residual peroxide was measured at the manufacturers minimum recommended storage time (6 hours for Clear Care Plus and 4 hours for PeroxiClear).
Time Frame: Day 30, each product
Population: Intention to treat participants with non-missing observations
Measure: Mean (Standard Deviation); unit: parts per million (ppm)
Units Other Than Participants: Lens Cases
Groups:
- PeroxiClear: PeroxiClear Lens Cases
- Clear Care Plus: Clear Care Plus Lens Cases
Arm/Group | PeroxiClear | Clear Care Plus
Number analyzed (Participants) | 132 | 132
Number analyzed (Lens Cases) | 130 | 130
parts per million (ppm) | 229.7 (280.13) | 26.2 (41.17)

2. Secondary Outcome: Mean Osmolality in Lens Cases at Day 30
Description: The used lens case was collected after approximately 30 days of use. Remaining liquid was removed and dry cases were shipped to a lab for analysis. 10 mL of the appropriate solution was added to each collected case. Osmolality was measured at the manufacturers minimum recommended storage time (6 hours for Clear Care Plus and 4 hours for PeroxiClear).
Time Frame: Day 30, each product
Population: Intention to treat participants with non-missing observations
Measure: Mean (Standard Deviation); unit: milliosmoles/kg (mOsm/kg)
Units Other Than Participants: Lens Cases
Arm/Group | PeroxiClear | Clear Care Plus
Number analyzed (Participants) | 132 | 132
Number analyzed (Lens Cases) | 130 | 130
milliosmoles/kg (mOsm/kg) | 345.1 (11.76) | 299.2 (7.63)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study from the signing of informed consent (up to 60 [+10] days).
Description: AEs were defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs, whether or not related to the medical device, obtained through solicited and spontaneous comments from all exposed participants and reported based on the treatment received. Ocular AEs are presented for both eyes combined.
Groups:
- PeroxiClear: While using PeroxiClear
- Clear Care Plus: While using Clear Care Plus
Arm/Group | PeroxiClear | Clear Care Plus
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/130
Other Adverse Events (participants affected / at risk) | 0/130 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.